CLINICAL TRIAL: NCT00162136
Title: Phase I Study of Ixabepilone Administered as a 24-Hour Infusion in Patients With Advanced Solid Malignancies
Brief Title: Clinical Study of Ixabepilone Administered as a 24 Hour Infusion in Patients With Solid Malignancies.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-085
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Results first posted 2010-01-27 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2016-02

CONDITIONS: Solid Malignancies
MeSH Terms: interventions — ixabepilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A1 (Experimental)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Intravenous (IV) Infusion; 10, 20, 30, 35, 40 & 45 mg/m2, once every 21 days (1 cycle), up to 9 cycles
  Other Names: IXEMPRA®

SUMMARY:
The purpose of this study is to determine the dose limiting toxicities, minimum tolerated dose and recommended dose for Phase II studies.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of a primary solid tumor
* measurable or non-measurable disease
* progressive disease
* men and women greater or equal to 18 years of age.

Exclusion Criteria:

* women of child bearing potential who are not using birth control
* women who are pregnant or breast feeding
* women with a positive pregnancy test on enrollment
* patients with brain metastasis
* prior treatment with Ixabepilone
* known history of human immunodeficiency virus (HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (3):
  - University Of Maryland, Baltimore, Maryland
  - The Cancer Institute Of New Jersey, New Brunswick, New Jersey
  - Cleveland Clinic Foundation, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 39 participants enrolled and 4 participants were never treated (2 reported serious adverse events [SAEs] prior to the first dose of study medication and were never treated; 1 had rapid decline in performance status and died prior to the first dose of study medication; no reason was given for the remaining participant).
Period: Overall Study
Arm/Group | Ixabepilone
Started | 35
Completed | 0 (Number of Participants still on treatment at study termination)
Not Completed | 35
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Disease Progression/Relapse | 23
Not completed — Investigator Request | 5
Not completed — Study Drug Toxicity | 4
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- 10 mg/m2; 20 mg/m2; 30 mg/m2; 35 mg/m2; 40 mg/m2; 45 mg/m2: Ixabepilone
- Total: Total of all reporting groups
Arm/Group | 10 mg/m2 | 20 mg/m2 | 30 mg/m2 | 35 mg/m2 | 40 mg/m2 | 45 mg/m2 | Total
Number analyzed (Participants) | 4 | 3 | 8 | 4 | 11 | 5 | 35
Age, Continuous [Mean (Full Range); unit: years] | 63.5 [54 to 74] | 59.0 [58 to 64] | 61.5 [39 to 70] | 59.5 [53 to 62] | 58.0 [53 to 79] | 52.0 [40 to 60] | 59.0 [39 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 5 | 2 | 5 | 3 | 16
  Male | 3 | 3 | 3 | 2 | 6 | 2 | 19
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 2 | 7 | 3 | 9 | 2 | 26
  Black | 0 | 1 | 0 | 1 | 1 | 2 | 5
  Asian | 1 | 0 | 1 | 0 | 1 | 1 | 4
Karnofsky Performance Status [Number; unit: participants] — The Karnofsky Performance Status (KPS) measures the ability of cancer patients to perform ordinary tasks. Scores are reported in multiples of 10 and range from 0 to 100; a higher score means the patient is better able to carry out daily activities.
  participants
    90 to 100 | 2 | 2 | 6 | 2 | 7 | 3 | 22
    70 to 80 | 2 | 1 | 2 | 2 | 4 | 2 | 13
    0 to 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities at Dose Level
Description: Dose limiting toxicities=any of the following events attributed to Ixabepilone occuring during the first cycle: grade 3/4 nausea, vomiting, or diarrhea despite medical intervention and/or prophylaxis; other Grade ≥3 nonhematological toxicity; any toxicity requiring study therapy discontinuation; delayed recovery from study therapy-related toxicity which delays scheduled re-treatment for >14 days; Grade 4 neutropenia for ≥5 consecutive days; grade 3/4 neutropenia with sepsis or a fever ≥38.5 C; thrombocytopenia <25,000 cells/mm3 or bleeding requiring a platelet transfusion.
Time Frame: Measures taken at Cycle 01 (21-day cycle)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | 10 mg/m2 | 20 mg/m2 | 30 mg/m2 | 35 mg/m2 | 40 mg/m2 | 45 mg/m2
Number analyzed (Participants) | 4 | 3 | 8 | 4 | 11 | 5
participants | 0 | 0 | 0 | 0 | 1 | 2

2. Secondary Outcome: Treatment Related Adverse Events (AEs), Serious Adverse Events (SAEs), Deaths, and AEs Leading to Discontinuation
Description: Adverse events (AEs) and Serious AEs (SAEs) considered possibly, probably, or certainly related to study treatment, graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death).
Time Frame: From time of screening through post study follow-up at a maximum of 21 9-day cycles. Toxicity assessments occured at least every 4 weeks until all study drug related toxicities.
Measure: Number; unit: Participants
Groups:
- Grade 1/2: Grade 1=Mild, Grade 2=Moderate
- Grade 3/4: Grade 3=Severe, Grade 4=Life-threatening or disabling
- All Grades: Grades 1-4
Arm/Group | Grade 1/2 | Grade 3/4 | All Grades
Number analyzed (Participants) | 35 | 35 | 35
Participants
  Any Treatment-Related AE | 12 | 21 | 33
  Nausea | 16 | 0 | 16
  Fatigue | 14 | 2 | 16
  Alopecia | 12 | 0 | 12
  Diarrhea | 11 | 0 | 11
  Peripheral sensory neuropathy | 9 | 0 | 9
  Stomatitis | 9 | 0 | 9
  Any SAE | 0 | 16 | 16
  Death within 30 days of last dose | 0 | 1 | 1
  Any AE leading to discontinuation | 0 | 5 | 5

3. Secondary Outcome: Hematology Results - Worst On-Study Grade
Description: Worst on-study grade based on laboratory values graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. (Grade 1=Mild, Grade 2=Moderate, Grade 3=Severe, Grade 4=Life-threatening or disabling, Grade 5=Death).
Time Frame: Baseline (within 2 weeks of dosing), weekly, and within 72 hours prior to each subsequent 21-day cycle. If CTC Grade 4 hematologic toxicity is observed, complete blood count plus differential and platelets repeated every 3 days until resolution.
Measure: Number; unit: Participants
Groups:
- Grade 0: Absent
- Grade 1: Mild
- Grade 2: Moderate
- Grade 3: Severe
- Grade 4: Life-threatening or disabling
Arm/Group | Grade 0 | Grade 1 | Grade 2 | Grade 3 | Grade 4
Number analyzed (Participants) | 35 | 35 | 35 | 35 | 35
Participants
  White Blood Cells | 5 | 5 | 8 | 10 | 7
  Absolute Neutrophil Count | 8 | 5 | 6 | 5 | 11
  Hemoglobin | 1 | 14 | 13 | 7 | 0
  Platelets | 21 | 9 | 0 | 3 | 2

4. Secondary Outcome: Mean Plasma Concentration of Ixabepilone at 40 mg/m2 Dose Level
Description: Mean concentrations over full time period for the 40 mg/mg2 dose level, established as the Maximum Tolerated Dose. (The Maximum Tolerated Dose was established as 40 mg/m2, based on an investiagtion of Dose Limiting Toxicities, which consisted of Febrile Neutropenia (at 40 mg/m2) in 1 participant and Grade 4 neutropenia lasting ≥5 days (at 45 mg/m2)in 2 participants.)
Time Frame: through 72 hours after start of infusion
Population: All participants treated at the 40 mg/m2 dose level.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treated Subjects: All treated subjects with measurement at timepoint
Arm/Group | Treated Subjects
Number analyzed (Participants) | 11
ng/mL
  Hour 0.00 (n=11) | 0 (0)
  Hour 1.00 (n=11) | 20.79 (14.12)
  Hour 2.00 (n=11) | 24.31 (13.64)
  Hour 4.00 (n=11) | 33.15 (32.75)
  Hour 8.00 (n=11) | 32.04 (16.20)
  Hour 12.00 (n=11) | 35.25 (11.96)
  Hour 16.00 (n=11) | 44.47 (13.80)
  Hour 20.00 (n=11) | 55.05 (29.41)
  Hour 24.00 (n=11) | 54.71 (23.63)
  Hour 25.00 (n=10) | 35.59 (24.51)
  Hour 26.00 (n=10) | 33.70 (17.17)
  Hour 27.00 (n=10) | 35.15 (20.47)
  Hour 72.00 (n=10) | 27.45 (47.71)

5. Secondary Outcome: Best Tumor Response, According to Response Evaluation Criteria in Solid Tumors (RECIST)
Description: RECIST criteria, wherein complete response = disappearance of all target lesions; partial response = 30% decrease in the sum of the longest diameter of target lesions; progressive disease = 20% increase in the sum of the longest diameter of target lesions, and stable disease = small changes that do not meet above criteria.
Time Frame: At Baseline (up to 2 weeks prior to starting therapy), after every 2nd cycle, and at post study follow-upn after a maximum of 9 cycles.
Measure: Number; unit: Participants
Arm/Group | All Treated Participants
Number analyzed (Participants) | 35
Participants
  Complete Response | 0
  Partial Response | 0
  Stable Disease | 14
  Progressive Disease | 15
  Unable to Determine | 6

ADVERSE EVENTS:
Arm/Group | Ixa 10 mg/m2 | Ixa 20 mg/m2 | Ixa 30 mg/m2 | Ixa 35 mg/m2 | Ixa 40 mg/m2 | Ixa 45 mg/m2
Serious Adverse Events (participants affected / at risk) | 2/4 | 2/3 | 4/8 | 1/4 | 5/11 | 2/5
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 8/8 | 4/4 | 11/11 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixa 10 mg/m2 (N=4) | Ixa 20 mg/m2 (N=3) | Ixa 30 mg/m2 (N=8) | Ixa 35 mg/m2 (N=4) | Ixa 40 mg/m2 (N=11) | Ixa 45 mg/m2 (N=5)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
HEPATORENAL SYNDROME (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
HEMIPARESIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
ILEUS (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
UROSEPSIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
SEPTIC SHOCK (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
GLUCOSE TOLERANCE IMPAIRED (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 1 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
TRACHEO-OESOPHAGEAL FISTULA (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
FATIGUE (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixa 10 mg/m2 (N=4) | Ixa 20 mg/m2 (N=3) | Ixa 30 mg/m2 (N=8) | Ixa 35 mg/m2 (N=4) | Ixa 40 mg/m2 (N=11) | Ixa 45 mg/m2 (N=5)
DRY EYE (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
ECTROPION (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
PHOTOPSIA (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 1
EYE OEDEMA (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
EYE IRRITATION (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
VISION BLURRED (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
ERYTHEMA OF EYELID (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 1 | 4 | 1 | 1 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 2
URINE OUTPUT DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
BLOOD ALBUMIN DECREASED (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
BLOOD CALCIUM DECREASED (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
PLATELET COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
BLOOD PHOSPHORUS DECREASED (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
GASTRIC OCCULT BLOOD POSITIVE (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
WAIST CIRCUMFERENCE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 0 | 1 | 0 | 1 | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 | 0 | 1 | 0 | 1 | 0
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
FLUSHING (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 0
HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0 | 2 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 1 | 0 | 0 | 0
ANXIETY (Psychiatric disorders) | 0 | 1 | 2 | 0 | 2 | 0
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2 | 0
AGITATION (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
NIGHTMARE (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 1
ABNORMAL DREAMS (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 0
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 2
TREMOR (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 1
APHASIA (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
HEADACHE (Nervous system disorders) | 1 | 1 | 3 | 1 | 0 | 2
DIZZINESS (Nervous system disorders) | 0 | 2 | 1 | 0 | 2 | 0
DYSGEUSIA (Nervous system disorders) | 0 | 2 | 3 | 1 | 1 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 0
HYPOAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
MENTAL IMPAIRMENT (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
SYNCOPE VASOVAGAL (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 | 1 | 3 | 1 | 5 | 1
NAUSEA (Gastrointestinal disorders) | 2 | 3 | 7 | 2 | 6 | 0
LIP DRY (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
RETCHING (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 2 | 4 | 0 | 3 | 0
CHEILITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 5 | 3 | 6 | 0
DRY MOUTH (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 3 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
DYSPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GLOSSITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
ORAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
TOOTHACHE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
STOMATITIS (Gastrointestinal disorders) | 0 | 1 | 3 | 0 | 4 | 1
LOOSE TOOTH (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
ODYNOPHAGIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 2 | 4 | 1 | 5 | 2
OESOPHAGITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 3 | 0 | 2 | 0
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
GINGIVAL ERYTHEMA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
STOMACH DISCOMFORT (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 0
TONGUE DISCOLOURATION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPOACUSIS (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
RHINITIS (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
CANDIDIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
TINEA PEDIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
FOLLICULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
TOOTH INFECTION (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
ORAL CANDIDIASIS (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
NOCTURIA (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
POLLAKIURIA (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1
RENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
ACUTE PRERENAL FAILURE (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
STRESS URINARY INCONTINENCE (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0
ANOREXIA (Metabolism and nutrition disorders) | 0 | 1 | 4 | 2 | 2 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 2 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | 0
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 1 | 1 | 5 | 2
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 4 | 1 | 7 | 3
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 4 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 6 | 1 | 5 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 2 | 0
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
SKIN DISORDER (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
SUBCUTANEOUS NODULE (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
ANIMAL BITE (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 4 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 4 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 3 | 1
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
JOINT STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 3 | 0
MOBILITY DECREASED (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
SENSATION OF HEAVINESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 4 | 2 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1 | 2 | 1
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0
PHARYNGOLARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 0
PAIN (General disorders) | 0 | 1 | 0 | 1 | 1 | 0
CHILLS (General disorders) | 2 | 2 | 0 | 0 | 1 | 1
THIRST (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
FATIGUE (General disorders) | 1 | 3 | 6 | 3 | 8 | 3
PYREXIA (General disorders) | 0 | 0 | 2 | 2 | 2 | 0
ASTHENIA (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
FEELING COLD (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 1 | 2 | 0 | 1 | 0
MUCOSAL HAEMORRHAGE (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 0 | 0 | 2 | 0 | 2 | 1
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
CATHETER RELATED COMPLICATION (General disorders) | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.